CLINICAL TRIAL: NCT03109626
Title: Translating Molecular Pathology Into a Therapeutic Strategy in SCA38, a Newly Identified Form of Spinocerebellar Ataxia
Brief Title: Docosahexaenoic Acid (DHA) Replacement for Treatment in Spinocerebellar Ataxia 38
Acronym: SCA38DHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Borroni (Other)
Responsible Party: Sponsor-Investigator, Barbara Borroni, Associated Professor of Neurology, MD, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Organization: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CE NP1821
Record Dates: First submitted 2017-03-31; First posted 2017-04-12 (Actual); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: SCA38
Keywords: DHA, replacement, treatment, brain PET-FDG, ataxia
MeSH Terms: conditions — Ataxia

STUDY DESIGN:
Intervention Model Description: double-blind randomised placebo-controlled phase, followed by an open-label phase
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DHA administration (Active Comparator): DHA 600 mg/day will be administered for 16 weeks to 5 patients in double blind
  Interventions: Dietary Supplement: DHA
- placebo administration (Placebo Comparator): placebo will be made with the same colour and taste, in softgel as DHA, and will be administered for 16 weeks to 5 patients in double blind.
  Interventions: Dietary Supplement: DHA

INTERVENTIONS:
Dietary Supplement: DHA

SUMMARY:
The project will study a therapeutic approach in Spinocerebellar Ataxia (SCA38) by DHA replacement. SCA38 is caused by missense mutations in the ELOVL5 (Elongation of very long chain fatty acids protein 5) gene.

Background/Rationale: ELOVL5 is a microsomal fatty acid elongase gene required for the synthesis of arachidonic acid and DHA. In brain, it shows a peculiar high expression in cerebellar Purkinje cells.

The ELOVL5 products, such as DHA, are decreased in SCA38 patients serum and DHA administered as a dietary supplement has been shown to improve SARA scores, to ameliorate quality of life, and to increase brain cerebellar hypometabolism (FDG-PET) in two SCA38 patients.

Experimental Plan: The investigators will perform a randomized placebo-controlled trial by DHA supplementation on ten SCA38 patients, followed by an open-label phase.

Expected results: DHA supplementation should be able to improve symptoms in SCA38 and to improve cerebellar hypometabolism in these patients.

DETAILED DESCRIPTION:
Spinocerebellar ataxias (SCAs) include over thirty different subtypes of central nervous system diseases that affect approximately 1 in 30,000 persons. The investigators have identified the causative gene for SCA38, a novel rare form of cerebellar ataxia. Estimated frequency of the disease is below 1% of SCAs. The disease gene encodes an enzyme involved in omega-3 fatty acid biosynthesis, whose products are reduced in SCA38 patients' serum.

The investigators reasoned that the administration of specific omega-3 fatty acids could ameliorate the disease symptoms in SCA38 patients. Indeed, preliminary data obtained in a pilot trial on two patients, now in their 8th-month therapy, are remarkable, with an improvement of disease symptoms and quality of life, without any adverse effect.

The investigators will perform a clinical trial to prove this therapeutic strategy of SCA38. The investigators will evaluate clinical SARA scores, ICARS scores, brain PET images, and plasma metabolic pattern in ten SCA38 patients.

The trial will consist of two phases: 1) a randomized double-blind placebo/treatment (600 mg DHA/day) from T0 (baseline observation) to T1 (evaluation at four-month). Patients who will meet the study eligibility criteria will be randomized to receive the drug or the placebo (ratio 1:1). A second open-label phase on all patients from T2 (6 months) to T5 (30 months) will be performed with repeated measures of the medication group (n=10).

Patients will complete a personal diary during the whole treatment and a quality of life questionnaire at each visit. The primary outcome will be the clinical improvement, whilst secondary outcome will be considered the improvement of brain metabolism by PET-FDG.

At each time point, clinical evaluation (video-record of SARA/ICARS scores) will be performed. Videos will be randomized and evaluated blindly by two independently clinicians.

At T0, T1, T2, T5, patients will undergo brain PET-FDG scan. PET-FDG scans will be performed by the same scanner at the University of Brescia.

This project will provide helpful data on possible replacement treatment in this novel form of cerebellar degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Mutations p.Gly230Val in ELOVL5 gene
* Clinical symptoms of ataxia

Exclusion Criteria:

* Use of fish oil or DHA dietary supplement within 30 days prior the enrollment in the present trial
* Evidence of poorly controlled diabetes (defined as hemoglobin A1c > 8% in patients with diabetes)
* Average alcohol consumption of more than one drink or equivalent (>12 g) per day or more than two drinks on any 1 day over the 30 days prior to screening.
* Serum creatinine level 2.0 mg/dL or greater or currently on dialysis
* Evidence of drug abuse within 6 months prior to entering the study or during the screening period
* Reported poor compliance to drug assumption
* Bedridden patients (SARA score >23)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-06-17 (Actual); Primary Completion 2015-09-17 (Actual); Study Completion 2018-06-25 (Actual)

PRIMARY OUTCOMES:
Change from Baseline SARA score at 16 weeks and 40 weeks | baseline, 16 weeks, 40 weeks
  improvement of ataxia by SARA scores
Change from Baseline ICARS score at 16 weeks and 40 weeks | baseline, 16 weeks, 40 weeks
  improvement of ataxia by ICARS scores

SECONDARY OUTCOMES:
Brain FDG-PET | baseline, 16 weeks, 40 weeks
  improvement of cerebellar hypometabolism

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Borroni, MD, Principal Investigator — AO Spedali Civili
Locations (1):
- AO Spedali Civili, Brescia, BS, Italy

IPD SHARING:
Plan to Share IPD: Yes
to share data after study publication

REFERENCES:
- [Background] Di Gregorio E, Borroni B, Giorgio E, Lacerenza D, Ferrero M, Lo Buono N, Ragusa N, Mancini C, Gaussen M, Calcia A, Mitro N, Hoxha E, Mura I, Coviello DA, Moon YA, Tesson C, Vaula G, Couarch P, Orsi L, Duregon E, Papotti MG, Deleuze JF, Imbert J, Costanzi C, Padovani A, Giunti P, Maillet-Vioud M, Durr A, Brice A, Tempia F, Funaro A, Boccone L, Caruso D, Stevanin G, Brusco A. ELOVL5 mutations cause spinocerebellar ataxia 38. Am J Hum Genet. 2014 Aug 7;95(2):209-17. doi: 10.1016/j.ajhg.2014.07.001. Epub 2014 Jul 24. PMID 25065913